CLINICAL TRIAL: NCT02236858
Title: Clinical Trial of Air Cleaners to Improve Indoor Air Quality and COPD Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NA_00085617; 1R01ES022607 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-09-11 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham HEPA Air Cleaner (Sham Comparator): Sham HEPA Air Cleaner and Delayed Intervention. Homes in the control group will receive sham air cleaners that have the internal HEPA and carbon filters removed, but which will run normally, including similar noise, airflow and overall appearance compared to active air cleaners, thus blinding participants to filter status.
  Interventions: Device: Sham HEPA Air Cleaner
- HEPA Air Cleaner (Active Comparator): HEPA Air Cleaner also containing carbon filters (Austin HealthMate HM400) and capable of removing PM and NO2 will be placed in the bedroom and room where the participant reports spending the most time. These air cleaners are suitably sized to provide clean air delivery rates for the rooms in which they will be placed. Participants will be instructed to run the air cleaners continually during the course of the study and the units will be modified to prevent them from being turned off by the participants.
  Interventions: Device: HEPA Air Cleaner

INTERVENTIONS:
Device: HEPA Air Cleaner — Air cleaners containing HEPA and carbon filters (Austin HealthMate HM400) and capable of removing PM and NO2 will be placed in the bedroom and room where the participant reports spending the most time.
  Arms: HEPA Air Cleaner
Device: Sham HEPA Air Cleaner — Homes in the control group will receive sham air cleaners that have the internal HEPA and carbon filters removed, but which will run normally, including similar noise, airflow and overall appearance compared to active air cleaners, thus blinding participants to filter status.
  Arms: Sham HEPA Air Cleaner

SUMMARY:
Objectives (include all primary and secondary objectives)

Specific Aim #1: To determine whether an air cleaner intervention to improve home air quality will improve respiratory symptoms, quality of life, lung function and reduce risk of exacerbations in former smokers with COPD.

Hypothesis: An intervention using high-efficiency particulate air (HEPA) and carbon filter air cleaners in homes of former smokers with COPD will improve respiratory symptoms, quality of life, and lung function and reduce risk of COPD exacerbations compared with placebo (sham air cleaners).

Specific Aim #2: To determine whether an air cleaner intervention to improve home air quality will be associated with intermediate outcome measures known to be linked with long term outcomes in COPD, including airway and systemic markers of inflammation and oxidative stress, in former smokers with COPD.

Hypothesis 2: An intervention using HEPA and carbon filter air cleaners in homes of formers smokers with COPD will be associated with lower levels of markers of inflammation and oxidative stress known to be associated with adverse outcomes in patients with COPD.

DETAILED DESCRIPTION:
This research is being done to learn whether an air cleaner intervention to improve home air quality (particulate matter (PM) and nitrogen dioxide (NO2) reduction) will improve respiratory symptoms, quality of life, lung function, and reduce risk of exacerbations in former smokers with COPD.

The investigators will place air pollution monitors in the home to measure the air quality over five 1-week periods (at 3 month and 1 week pre-intervention, and 1 week, 3 months and 6 months post-intervention). During each week of monitoring, the investigators will ask that a diary be kept of breathing and how the participants are feeling every day.

Participant will have 5 home visits and 5 clinic visits and monthly telephone calls during this time to see how the participant is feeling. One week after each home visit, the monitoring equipment will be picked up. After the 2nd monitoring period, active or sham air cleaners will be placed in home.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years,
* Physician diagnosis of COPD,
* Global Initiative for Obstructive Lung Disease (GOLD) Stage II-IV disease with Forced Expiratory Volume (FEV1)/ Forced Vital Capacity (FVC) ≤70% and FEV1 (% predicted) <80%,
* Tobacco exposure ≥ 10 pack-years, and
* Former smoker. We will employ a combination of self-report and a biochemical marker to identify former-smokers. Exhaled CO (eCO) will be used as a marker of smoking status, as it is easy to perform, provides immediate data and is non-invasive. Former-smokers will be those who report no current smoking in the past 1 year AND have exhaled CO levels ≤ 6ppm. This threshold was chosen to maximize the chance of distinguishing true smokers and ex-smokers (>95%).

Exclusion Criteria:

* Chronic systemic corticosteroids (≥ 3 months continuous use in past 12 months),
* Other chronic lung disease including asthma,
* Living in location other than home (e.g., long term care facility) and
* Home owner or home occupant planning to move or change residence within the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Change from baseline and at 6 months post randomization
  St. George's Respiratory Questionnaire (SGRQ). The total score is from 0 to 100. Higher scores indicate more limitations

SECONDARY OUTCOMES:
Health care utilization | Baseline through end of study (approximately 6 months post-randomization)
  Aggregate Exacerbations including (need for oral corticosteroids or antibiotics for worsening respiratory symptoms, emergency department (ED) visit or hospitalization).
  During this 6 months exacerbations will be collected at monthly telephone calls and at 3 and 6 month clinic visits. Whether an exacerbation occurred over this 6 month period will be assessed.
Change in Dyspnea (mMRC) | Change from baseline and 3 months post-randomization
  Dyspnea will be assessed using the modified medical research Council questionnaire (mMRC). The total score is from 0 (no dyspnea) to 2 (severe dyspnea).
Change in Dyspnea (mMRC) | Change from baseline and 6 months post-randomization
  Dyspnea will be assessed using the modified medical research Council questionnaire (mMRC). The total score is from 0 (no dyspnea) to 2 (severe dyspnea).
Change in COPD health status | Change from baseline and 3 months post randomization
  Functional status will be assessed with the COPD assessment test (CAT). The total score is from 0 to 40. Higher scores indicate worse COPD control
Change in COPD health status | Change from baseline and 6 months post randomization
  Functional status will be assessed with the COPD assessment test (CAT). The total score is from 0 to 40. Higher scores indicate worse COPD control
Change in Functional status | Change from baseline and 3 months post randomization
  Functional status will be assessed with the 6 minute walk test. We will assess the distance (in meters) covered a time of 6 minutes.
Change in Functional status | Change from baseline and 6 months post randomization
  Functional status will be assessed with the 6 minute walk test. We will assess the distance (in meters) covered a time of 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N Hansel, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Woo H, Koehler K, Putcha N, Lorizio W, McCormack M, Peng R, Hansel NN. Principal stratification analysis to determine health benefit of indoor air pollution reduction in a randomized environmental intervention in COPD: Results from the CLEAN AIR study. Sci Total Environ. 2023 Apr 10;868:161573. doi: 10.1016/j.scitotenv.2023.161573. Epub 2023 Jan 18. PMID 36669663